CLINICAL TRIAL: NCT07294976
Title: Evaluation of Actual Maximum Gain in Bone Anchored Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BC126
Record Dates: First submitted 2025-11-27; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All study participants (Experimental): All study patients will sequentially be measured with Device A, Device B and Device C
  Interventions: Device: Bone Anchored Device A; Device: Bone Anchored Device B; Device: Bone Anchored Device C

INTERVENTIONS:
Device: Bone Anchored Device A — Fitting Device A
Device: Bone Anchored Device B — Fitting Device B
Device: Bone Anchored Device C — Fitting Device C

SUMMARY:
This study will look at how much sound amplification (gain) different bone-anchored hearing devices can provide. The goal is to understand if there are differences between devices and whether these differences affect how well the devices meet the hearing needs of users.

Bone-anchored hearing systems send sound vibrations directly to the inner ear through a small implant in the skull. The amount of amplification a device can provide is important for people with hearing loss. However, the actual maximum amplification available to a user depends on feedback control during fitting and can vary between devices and individuals.

In this study, the actual maximum amplification of Device A and Device B will be compared. In addition the actual maximum amplification of Device A will be compared to Device C as well as the Device B compared to Device C. It will also be investigated whether the amplification limits the prescribed settings for the users.

ELIGIBILITY:
Inclusion Criteria:

1. BAHS user with an Oticon Medical compatible abutment
2. Signed Informed Consent Form
3. Adult, 18 years or older
4. MHL with pure tone average (PTA) bone conduction (BC) threshold (measured at 0.5, 1, 2 and 3 kHz) of 25-65dB HL on the indicated ear
5. MHL with an air-bone-gap (difference between BC and AC thresholds) of at least 15 dB measured at 0.5, 1, 2 and 3 kHz
6. At least 3 months of experience using a bone conduction device.
7. Fluent in Swedish to be able to read and understand patient information and informed consent process

Exclusion Criteria:

1. Participation in another clinical investigation which might cause interference with study participation.
2. Subjects who do not have the ability or are unwilling to follow investigational procedures/requirements, e.g. to complete questionnaires, according to investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Difference in actual maximum gain in dB, between Device A compared to Device B for the mean average of the frequencies 500, 1000, 2000, 3000 and 4000 | Baseline, at fitting

SECONDARY OUTCOMES:
Difference in actual maximum gain in dB, between Device A compared to Device B for the for the mean average of the frequencies 500, 1000, 2000 and 4000 | Baseline, at fitting
Difference in actual maximum gain in dB, between Device A compared to Device B across frequencies 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 kHz | Baseline, at fitting
Difference in actual maximum gain in dB, between Device C compared to Device B for the mean average of the frequencies 500, 1000, 2000, 3000 and 4000 | Baseline, at fitting
Difference in actual maximum gain in dB, between Device C compared to Device B for the mean average of the frequencies 500, 1000, 2000 and 4000 | Baseline, at fitting
Difference in actual maximum gain in dB, between Device C compared to Device B across frequencies 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 kHz | Baseline, at fitting
Number of subjects with a limitation of the prescribed gain in any frequency band with Device A, Device B and Device C | Baseline, at fitting

CONTACTS AND LOCATIONS:
Locations (1):
- Göteborgs Universitet, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No